CLINICAL TRIAL: NCT00250653
Title: A Fifty-two-week, Multicenter, Open-label Study Evaluating the Long-term Safety and Tolerability of Saredutant in Adult and Elderly Patients With Major Depressive Disorder
Brief Title: A Fifty-two-week Study to Evaluate the Safety of Saredutant in Adult and Elderly Patients With Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LTS5577; Saredutant (SR48968C)
Record Dates: First submitted 2005-11-07; First posted 2005-11-08 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2012-02

CONDITIONS: Depressive Disorder
Keywords: depression; antidepressive agents; clinical trial
MeSH Terms: conditions — Depressive Disorder; Depression | interventions — SR 48968

INTERVENTIONS:
Drug: Saredutant succinate (SR48968C)

SUMMARY:
The purpose of the study is to evaluate the long-term safety of saredutant (or SR48968C) in adult and elderly patients with depression.The primary objective is to evaluate the long-term safety and tolerability of a 100 mg dose of saredutant in adult and elderly patients with depression. The secondary objective is to evaluate blood levels of saredutant.

DETAILED DESCRIPTION:
The study is a multicenter, US, open-label study consisting of two segments (A and B). Segment A is a minimum 1-week (maximum 4-week) screening period and Segment B is a 52-week, open-label period. All treated patients must complete a post-study telephone visit and a post-study office visit 3 days and 1 week, respectively, after intake of the last dose of study medication.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients.
* At least 18 years of age.
* Inpatients or outpatients.
* Written informed consent from the patient and/or legally authorized representative.
* Able to comply with the protocol and follow written and verbal instructions.
* Subjects of childbearing potential must have a confirmed negative serum b-hCG test prior to entry into Segment B and must employ an acceptable method of birth control (e.g., oral, depot, or implanted contraceptive method, IUDs, sterilization, barrier methods in conjunction with spermicide).
* Diagnosis of major depressive disorder, as defined by Diagnostic and Statistical Manual of Mental Disorders, 4th edition, Text Revision criteria and confirmed by the semi-structured Mini International Neuropsychiatric Interview (MINI), recurrent episode for at least one month prior to the entry.
* Minimum total score of 18 on the Hamilton Depression Rating Scale (HAM-D).

Exclusion Criteria:

* Patients whose current depressive episode is diagnosed with psychotic features, catatonic features, seasonal pattern or post-partum onset.
* The duration of the current depressive episode is greater than 2 years.
* Patients who are currently suicidal or have a history of a suicide attempt within 3 years prior to entry.
* Patients whose current depressive episode is secondary to a general medical disorder.
* Patients with a history or presence of bipolar disorders or psychotic disorders according to the D and L criteria of the MINI.
* Patients with alcohol dependence or abuse or substance dependence or abuse in the past 12 months except nicotine or caffeine dependence.
* Patients with a history of failure to respond to treatment with paroxetine or other antidepressant medications.
* Patients who have used the following prior to entry into Segment B: fluoxetine within 28 days, any monoamine oxidase inhibitor within 21 days, any other antidepressant, anxiolytic, sedative-hypnotic, or mood-stabilizer (lithium, anticonvulsants) within 7 days except permitted concomitant medications.
* Females who are pregnant or breast-feeding.
* Severe or unstable cardiovascular, renal, hepatic, respiratory, hematological, endocrinological, neurological, or other somatic disease that might interfere with the evaluation of study medication.
* History of seizures other than a single childhood febrile seizure.
* ECG abnormalities of potential clinical significance including a QT interval with Bazett's correction of 500 msec or more at entry.
* Use of known inducers or potent inhibitors of CYP3A4 within 7 days of entry.
* Use of drugs with known risk for Torsade de Pointes within 7 days of entry into Segment B.
* Participation in a clinical trial of an experimental therapy within 30 days prior to entry or prior participation in a clinical trial of saredutant.
* Patients with a positive HbsAg or anti-HCV antibody test at screening.
* Patients with any of the following at screening: ALT >2 times the upper limit of the normal range (XULN), AST >2XULN, GGT >3XULN, total or conjugated bilirubin >ULN
* Elderly patients with a Mini-Mental State Examination total of score of <25.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 365 (Actual)
Dates: Start 2005-05; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the proportion of patients experiencing at least one treatment-emergent adverse event.

SECONDARY OUTCOMES:
The main secondary outcomes are incidences of potentially clinically significant abnormalities and the changes from baseline in the values for clinical laboratories, vital signs, and electrocardiogram parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Administrative Office, Bridgewater, New Jersey, United States